CLINICAL TRIAL: NCT00754065
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Group, 2-arm Study to Show Superiority of the Oral Contraceptive SH T00658ID Over Ortho Tri-Cyclen Lo on Hormone Withdrawal-associated Symptoms After 6 Cycles of Treatment.
Brief Title: To Compare SH T00658ID Over Ortho Tri-Cyclen Lo (US/Canada)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13108
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Contraception
Keywords: Oral contraceptive; Estradiol valerate and dienogest; EV/DNG; comparative tolerability
MeSH Terms: interventions — Estradiol; dienogest; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027) (Experimental): Daily oral administration of one capsule BAY86-5027 [estradiol valerate (EV) / dienogest (DNG)] for 26 days, followed by one capsule placebo for 2 days (28 days total per cycle) for 13 treatment cycles (treatment encapsulated)
  Interventions: Drug: Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027)
- Ortho Tri-Cyclen Lo (Active Comparator): Daily oral administration of one capsule Ortho Tri-Cyclen Lo [Ethinylestradiol (EE)/ Norgestimate (NGM)] for 21 days, followed by one capsule placebo for 7 days (28 days total per cycle) for 13 treatment cycles (treatment encapsulated)
  Interventions: Drug: Ortho Tri Cyclen Lo

INTERVENTIONS:
Drug: Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027) — Estradiol valerate (EV) and dienogest (DNG). Sequential 4-phasic regimen. Daily oral administration of one encapsulated BAY86-5027 for 28 days per Cycle, for 13 treatment cycles: Days 1-2, 3.0 mg EV; Days 3-7, 2.0 mg EV+2.0 mg DNG; Days 8-24, 2.0 mg EV+3.0 mg DNG; Days 25-26, 1.0 mg EV; Days 27-28, placebo
  Arms: Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027)
Drug: Ortho Tri Cyclen Lo — Dose--Ethinylestradiol (EE) + Norgestimate (NGM) Triphasic 21-day regimen. Daily oral administration of one encapsulated Ortho Tri-Cyclen Lo for 28 days per Cycle, for 13 treatment cycles: Days 1-7, 0.025 mg EE+0.180 NGM; Days 8-14, 0.025 mg EE+0.215 NGM; Days 15-21, 0.025 mg EE+0.250 NGM; Days 27-28, placebo
  Arms: Ortho Tri-Cyclen Lo

SUMMARY:
The objective of the study is to compare the oral contraceptive (OC) SH T00658ID over Ortho Tri-Cyclen Lo administered for 13 cycles to healthy female volunteers between 18 and 50 years of age who request oral contraceptive protection. Subjects on a levonorgestrel (LNG), norgestimate (NGM), norethindrone or norethindrone acetate containing oral contraceptive in a 21-day regimen suffering from hormone withdrawal-associated symptoms such as pelvic pain or headache or both, and willing to continue OC use but to switch to SH T00658ID or Ortho Tri-Cyclen Lo.

DETAILED DESCRIPTION:
Safety issues are addressed in the Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Age between 18 and 50 years (inclusive), smokers maximum age of 35 years (inclusive) at Visit 1
* Otherwise healthy female subjects requesting contraception and currently using a LNG, NGM, or norethindrone/norethindrone acetate containing OC in a 21-day regimen and suffering from at least moderate pelvic pain, headache or both defined by an average of the highest 3 values of >/=35 mm on a VAS during cycle days 22-28 (35 mm VAS is the expected standard deviation of the population VAS reduction)
* Normal or clinically insignificant cervical smear not requiring further follow up (a cervical smear has to be taken at screening visit or a normal result has to be documented within the last 6 months before screening) Women with atypical squamous cell of undetermined significance (ASCUS) can be included if they have a negative human papilloma virus (HPV) test result. The laboratory will perform an HPV test if the Pap smear result is ASCUS.
* Able to tolerate ibuprofen and willing to use only ibuprofen supplied by the investigator

Exclusion Criteria:

* Pregnancy or lactation (less than three cycles since delivery, abortion, or lactation before start of treatment)
* Body mass index (BMI) >32 kg/m2
* Hypersensitivity to any of the study drug ingredients
* Individuals not willing to consume pork and beef products. Women may be included if they are willing to take the capsules
* Safety relevant laboratory values, provided by the central laboratory, outside inclusion range before start of treatment
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study medication (such as but not limited to duodenal ulcers, gastritis, gastrectomy or gastric resection surgery, or renal compromise)
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Any disease or condition that may worsen under hormonal treatment
* Undiagnosed abnormal genital bleeding
* Abuse of alcohol, drugs, or medicines (eg, laxatives)
* Other contraceptive methods
* Any medication that could result in excessive accumulation, impaired metabolism, or altered excretion of the study drug or interfere with the conduct of the study or the interpretation of the results
* Simultaneous participation in another clinical trial prior to study entry that might have an impact on the study objectives at the discretion of the investigator
* Major surgery scheduled for the study period
* Subject is a dependent person, eg: a family member or member of the Investigator's staff
* Inability to cooperate with the study procedures for any reason, including language comprehension, psychiatric illness, inability to get to the study site

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 409 (Actual)
Dates: Start 2008-09-08 (Actual); Primary Completion 2011-05-10 (Actual); Study Completion 2011-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (53):
- United States (32):
  - Independence, Arizona
  - Phoenix, Arizona
  - Encinitas, California
  - San Diego, California
  - Santa Monica, California
  - Denver, Colorado
  - Littleton, Colorado
  - Clearwater, Florida
  - Jacksonville, Florida
  - West Palm Beach, Florida
  - Decatur, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Fishers, Indiana
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Metairie, Louisiana
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Bristol, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - Spokane, Washington
  - La Crosse, Wisconsin
- Canada (21):
  - Langley, British Columbia
  - Bathurst, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Corunna, Ontario
  - Downsview, Ontario
  - Hamilton, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Woodstock, Ontario
  - Charlottetown, Prince Edward Island
  - Drummondville, Quebec
  - Mirabel, Quebec
  - Pointe-Claire, Quebec
  - Shawinigan, Quebec
  - Ste-Foy, Quebec
  - Regina, Saskatchewan
  - Saskatoon, Saskatchewan
  - Québec

REFERENCES:
- [Result] Jensen JT, Parke S, Mellinger U, Serrani M, Mabey RG Jr. Hormone withdrawal-associated symptoms: comparison of oestradiol valerate/dienogest versus ethinylestradiol/norgestimate. Eur J Contracept Reprod Health Care. 2013 Aug;18(4):274-83. doi: 10.3109/13625187.2013.785516. Epub 2013 May 2. PMID 23638631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of first subject first visit was 08 Sep 2008. The date of last subject last visit was 10 May 2011.
Pre-assignment Details: A total of 776 participants were screened; 367 failed Screening, and 409 were randomized 1:1, of which 14 never received treatment, and 395 were treated (EV/DNG=191; EE/NGM=204). A total of 203 subjects (99 received EV/DNG and 104 EE/NGM) in the US and 192 (92 received EV/DNG and 100 EE/NGM) in Canada received at least one dose of the study drug.
Period: Overall Study
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Started | 203 | 206
Participants Received Treatment | 191 | 204
Cycle 6 | 141 | 153
Completed | 122 | 126
Not Completed | 81 | 80
Not completed — Never received treatment | 12 | 2
Not completed — Adverse Event | 19 | 25
Not completed — Lost to Follow-up | 7 | 11
Not completed — Protocol Violation | 12 | 10
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Pregnancy | 6 | 0
Not completed — Reason not specified or unknown, etc. | 21 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo | Total
Number analyzed (Participants) | 191 | 204 | 395
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.0 (6.6) | 26.5 (7.2) | 26.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 204 | 395
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 168 | 180 | 348
  Black | 9 | 9 | 18
  Hispanic | 6 | 10 | 16
  Asian | 4 | 2 | 6
  Other | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Change in Average of the 3 Highest Visual Analog Scale (VAS) Values of the Hormone Withdrawal-associated Symptoms Pelvic Pain or Headache During Cycle Days 22 to 28 From Baseline to Cycle 6
Description: Subject self-assessed pelvic pain or headache per visual analog scale (VAS) values during the menstrual/withdrawal bleeding episode and Baseline. The VAS consists of a 100 mm long straight line, with verbal anchors at either end, representing a continuum of pain intensity. Accordingly, the scale ranges from 0 mm (absence of pain) to 100 mm (unbearable pain), and the change ranges from -100 mm (best) to 100 mm (worst).
Time Frame: Day 22-28 from Baseline to Day 22-28 from Cycle 6 (28 days per Cycle)
Population: All participants in Full Analysis Set (FAS) with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 158 | 173
mm | 43.05 (23.58) | 34.97 (25.90)
Statistical Analysis 1: Comparison: Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) vs Ortho Tri-Cyclen Lo; 2-way ANOVA model with treatment and pain strata (headache and pelvic pain) as factors; Test type: Superiority or Other; p = 0.0024, ANOVA — Comparison of EV/DNG vs. EE/NGM; F-statistic = 9.3218

2. Secondary Outcome: The Change From Baseline to Cycle 6 in the Number of Ibuprofen Tablets Used as Rescue Medication
Description: Rescue medication use was standardized intake of 200 mg Ibuprofen tablets. Baseline period: 7 days (Day 22) before the first menstrual bleeding until Day 28 (normalized to a standard 28-day cycle). Treatment period: 7 days (Day 22) before the withdrawal bleeding (WB) of the 6th treatment cycle until Day 28 of the same cycle (normalized to a standard 28-day cycle). Number of tablets taken by each subject, and then the Mean and standard deviation (SD) derived.
Time Frame: From Baseline to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 148 | 157
Tablets
  Days 1-21 | -1.6 (9.9) | -3.0 (10.3)
  Days 22-28 | -5.8 (7.5) | -4.6 (8.0)

3. Secondary Outcome: The Change From Baseline to Cycle 13 in the Number of Ibuprofen Tablets Used as Rescue Medication
Description: Rescue medication use was standardized intake of 200 mg Ibuprofen tablets. Baseline period: 7 days (Day 22) before the first menstrual bleeding until Day 28 (normalized to a standard 28-day cycle). Treatment period: 7 days (Day 22) before the withdrawal bleeding (WB) of the 13th treatment cycle until Day 28 before the same cycle (normalized to a standard 28-day cycle). Number of tablets taken by each subject, and then the Mean and standard deviation ((SD) derived.
Time Frame: From Baseline to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 125 | 126
Tablets
  Days 1-21 | -2.3 (8.3) | -3.5 (12.0)
  Days 22-28 | -5.3 (7.6) | -5.2 (8.9)

4. Secondary Outcome: Change From Baseline to Cycle 6 in the Number of Days With at Least Moderate Pain/Intensity of Other Hormone-related Symptoms During Cycle Days 22-28
Description: Pain (pelvic, headache, bloating or swelling, breast tenderness, nausea or vomiting) during menstrual/withdrawal bleeding (WB) episode during cycle Days 22-28. Scores per day: 0 No pain; 1 Mild pain with no need for painkiller; 2 Moderate pain with need for painkiller; 3 Severe pain with need for painkiller. Baseline period: cycle Days 22-28 before 1st menstrual bleeding (normalized to a 7-day period). Treatment period: cycle Days 22-28 before WB of 6th treatment cycle until (normalized to a 7-day period). Score difference min -7 (best), max 7 (worst).
Time Frame: Day 22-28 from Baseline to Day 22-28 from Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 140 | 153
Days
  Headache | -1.950 (2.264) | -1.425 (2.223)
  Pelvic pain | -1.921 (2.219) | -1.830 (2.093)
  Bloating or swelling | -1.179 (2.051) | -1.131 (1.996)
  Breast tenderness | -0.536 (1.702) | -0.497 (1.755)
  Nausea or vomiting | -0.207 (1.089) | -0.229 (0.892)

5. Secondary Outcome: Change From Baseline to Cycle 13 in the Number of Days With at Least Moderate Pain/Intensity of Other Hormone-related Symptoms During Cycle Days 22-28
Description: Pain (pelvic, headache, bloating or swelling, breast tenderness, nausea or vomiting) during menstrual/withdrawal bleeding (WB) episode during cycle Days 22-28. Scores per day: 0 No pain; 1 Mild pain with no need for painkiller; 2 Moderate pain with need for painkiller; 3 Severe pain with need for painkiller. Baseline period: cycle Days 22-28 before 1st menstrual bleeding (normalized to a 7-day period). Treatment period: cycle Days 22-28 before WB of 13th treatment cycle (normalized to a 7-day period). Score difference min -7 (best), max 7 (worst).
Time Frame: Day 22-28 from Baseline to Day 22-28 from Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 121 | 124
Days
  Headache | -1.909 (2.317) | -1.419 (2.053)
  Pelvic pain | -2.091 (2.074) | -2.065 (2.233)
  Bloating or swelling | -0.959 (1.855) | -1.379 (1.868)
  Breast tenderness | -0.545 (1.727) | -0.677 (1.699)
  Nausea or vomiting | -0.248 (1.113) | -0.266 (1.148)

6. Secondary Outcome: Change From Baseline to Cycle 6 in the Number of Days With at Least Moderate Pain/Intensity of Individual Hormone-related Symptoms During Cycle Days 1-21
Description: Pain (pelvic, headache, bloating or swelling, breast tenderness, nausea or vomiting) during menstrual/withdrawal bleeding (WB) episode during cycle Days 1-21. Scores per day: 0 No pain; 1 Mild pain with no need for painkiller; 2 Moderate pain with need for painkiller; 3 Severe pain with need for painkiller. Baseline period: cycle Days 1-21 before 1st menstrual bleeding (normalized to a 21-day period). Treatment period: cycle Days 1-21 before WB of 6th treatment cycle (normalized to a 21-day period). Score difference min -21 (best), max 21 (worst).
Time Frame: Day 1-21 from Baseline to Day 1-21 from Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 143 | 157
Days
  Headache | -1.077 (3.407) | -0.968 (2.688)
  Pelvic pain | -0.399 (2.198) | -0.624 (2.147)
  Bloating or swelling | -0.531 (2.325) | -0.210 (2.056)
  Breast tenderness | -0.580 (1.798) | -0.248 (1.970)
  Nausea or vomiting | -0.182 (1.555) | -0.172 (1.507)

7. Secondary Outcome: Change From Baseline to Cycle 13 in the Number of Days With at Least Moderate Pain/Intensity of Individual Hormone-related Symptoms During Cycle Days 1-21
Description: Pain (pelvic, headache, bloating or swelling, breast tenderness, nausea or vomiting) during menstrual/withdrawal bleeding (WB) episode during cycle Days 1-21. Scores per day: 0 No pain; 1 Mild pain with no need for painkiller; 2 Moderate pain with need for painkiller; 3 Severe pain with need for painkiller. Baseline period: cycle Days 1-21 before 1st menstrual bleeding (normalized to a 21-day period). Treatment period: cycle Days 1-21 before WB of 13th treatment cycle (normalized to a 21-day period). Score difference min -21 (best), max 21 (worst).
Time Frame: Day 1-21 from Baseline to Day 1-21 from Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 129
Days
  Headache | -1.121 (3.122) | -0.767 (2.983)
  Pelvic pain | -0.274 (2.444) | -0.643 (2.113)
  Bloating or swelling | -0.492 (1.944) | -0.279 (2.140)
  Breast tenderness | -0.274 (1.467) | -0.217 (2.042)
  Nausea or vomiting | -0.298 (1.391) | -0.240 (1.457)

8. Secondary Outcome: Change From Baseline to Cycle 6 in the Number of Days With at Least Moderate Pain/Intensity of Individual Hormone-related Symptoms During the Hormone-free Interval Cycle Days 27 to 28 for EV/DNG and Cycle Days 22 to 28 for EE/NGM
Description: Pain (pelvic, headache, bloating or swelling, breast tenderness, nausea or vomiting) during menstrual/withdrawal bleeding (WB) episode (cycle Days 22-28). Scores per day: 0 No pain; 1 Mild pain with no need for painkiller; 2 Moderate pain with need for painkiller; 3 Severe pain with need for painkiller. Score difference min -2 (best), max 2 (worst) for the estradiol valerate (EV)/dienogest (DNG) group and min -7 (best), max 7 (worst) for the ethinylestradiol (EE)/norgestimate (NGM) group.
Time Frame: From Baseline to Cycle 6 (cycle Days 27 to 28 for EV/DNG and cycle Days 22 to 28 for EE/NGM, 28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 139 | 153
Days
  Headache | -0.424 (0.901) | -1.425 (2.223)
  Pelvic pain | -0.273 (1.013) | -1.830 (2.093)
  Bloating or swelling | -0.137 (0.773) | -1.131 (1.996)
  Breast tenderness | -0.043 (0.588) | -0.497 (1.755)
  Nausea or vomiting | -0.043 (0.378) | -0.229 (0.892)

9. Secondary Outcome: Change From Baseline to Cycle 13 in the Number of Days With at Least Moderate Pain/Intensity of Individual Hormone-related Symptoms During the Hormone-free Interval Cycle Days 27 to 28 for EV/DNG and Cycle Days 22 to 28 for EE/NGM
Description: Pain (pelvic, headache, bloating or swelling, breast tenderness, nausea or vomiting) during menstrual/withdrawal bleeding (WB) episode (cycle Days 22-28). Scores per day: 0 No pain; 1 Mild pain with no need for painkiller; 2 Moderate pain with need for painkiller; 3 Severe pain with need for painkiller. Score difference min -2 (best), max 2 (worst) for the EV/DNG group and min -7 (best), max 7 (worst) for the EE/NGM group.
Time Frame: From Baseline to Cycle 13 (cycle Days 27 to 28 for EV/DNG and cycle Days 22 to 28 for EE/NGM, 28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 121 | 124
Days
  Headache | -0.537 (0.904) | -1.419 (2.053)
  Pelvic pain | -0.322 (0.977) | -2.065 (2.233)
  Bloating or swelling | -0.107 (0.716) | -1.379 (1.868)
  Breast tenderness | -0.033 (0.515) | -0.677 (1.699)
  Nausea or vomiting | -0.033 (0.407) | -0.266 (1.148)

10. Secondary Outcome: Change From Baseline to Cycle 3 in the Average of the Three Highest VAS Values of the Hormone Withdrawal-associated Symptoms Pelvic Pain or Headache During Cycle Days 22 to 28
Description: as for outcome 1
Time Frame: Days 22-28 from Baseline to Days 22-28 from Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 154 | 171
mm | 36.92 (24.48) | 32.28 (25.77)

11. Secondary Outcome: Change From Baseline to Cycle 13 in the Average of the Three Highest VAS Values of the Hormone Withdrawal-associated Symptoms Pelvic Pain or Headache During Cycle Days 22 to 28
Description: as for outcome 1
Time Frame: Days 22-28 from Baseline to Days 22-28 from Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 122 | 126
mm | 45.89 (23.12) | 39.19 (27.68)

12. Secondary Outcome: Number of Days With Bleeding or Spotting in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment and includes the initial bleeding episode that triggered the first intake of study medication, meaning that the first treatment cycle includes 2 bleeding episodes.
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 164 | 180
Days | 19.0 (10.9) | 23.7 (8.2)

13. Secondary Outcome: Number of Days With Bleeding or Spotting in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 143 | 156
Days | 1.3 (9.2) | 18.8 (6.2)

14. Secondary Outcome: Number of Days With Bleeding or Spotting in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 132 | 138
Days | 14.1 (10.4) | 19.1 (6.5)

15. Secondary Outcome: Number of Days With Bleeding or Spotting in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 125 | 116
Days | 12.8 (9.1) | 19.4 (5.3)

16. Secondary Outcome: Number of Bleeding / Spotting Episodes in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment and includes the initial bleeding episode that triggered the first intake of study medication, meaning that the first treatment cycle includes 2 bleeding episodes. (Episode is a set of days with bleeding/spotting)
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 164 | 180
Episodes | 3.6 (1.4) | 3.7 (1.0)

17. Secondary Outcome: Number of Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment. (Episode is a set of days with bleeding/spotting)
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 143 | 156
Episodes | 3.3 (1.4) | 3.4 (0.9)

18. Secondary Outcome: Number of Bleeding / Spotting Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment. (Episode is a set of days with bleeding/spotting)
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 132 | 138
Episodes | 3.0 (1.4) | 3.3 (0.9)

19. Secondary Outcome: Number of Bleeding / Spotting Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment. (Episode is a set of days with bleeding/spotting)
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 125 | 116
Episodes | 3.0 (1.6) | 3.7 (0.8)

20. Secondary Outcome: Mean Length of Bleeding / Spotting Episodes in Reference Period 1
Description: as for outcome 12
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 160 | 180
Days | 4.82 (2.50) | 6.20 (2.22)

21. Secondary Outcome: Mean Length of Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 136 | 155
Days | 4.46 (2.31) | 5.71 (1.99)

22. Secondary Outcome: Mean Length of Bleeding / Spotting Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 122 | 138
Days | 4.70 (2.68) | 5.85 (1.53)

23. Secondary Outcome: Mean Length of Bleeding / Spotting Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 113 | 116
Days | 4.25 (1.57) | 5.65 (1.19)

24. Secondary Outcome: Maximum Length of Bleeding / Spotting Episodes in Reference Period 1
Description: as for outcome 12
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 160 | 180
Days | 7.8 (5.5) | 9.0 (4.3)

25. Secondary Outcome: Maximum Length of Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 136 | 155
Days | 6.2 (3.5) | 7.5 (3.7)

26. Secondary Outcome: Maximum Length of Bleeding / Spotting Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 122 | 138
Days | 6.2 (3.5) | 7.4 (2.8)

27. Secondary Outcome: Maximum Length of Bleeding / Spotting Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 113 | 116
Days | 5.7 (3.0) | 7.1 (2.3)

28. Secondary Outcome: Difference in Duration Between Longest and Shortest Bleeding / Spotting Episodes in Reference Period 1
Description: as for outcome 12
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 160 | 180
Days | 5.1 (5.3) | 5.1 (4.2)

29. Secondary Outcome: Difference in Duration Between Longest and Shortest Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 136 | 155
Days | 3.3 (3.2) | 3.5 (3.9)

30. Secondary Outcome: Difference in Duration Between Longest and Shortest Bleeding / Spotting Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 122 | 138
Days | 3.0 (3.0) | 3.1 (3.2)

31. Secondary Outcome: Difference in Duration Between Longest and Shortest Bleeding / Spotting Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 113 | 116
Days | 2.7 (3.3) | 2.8 (2.9)

32. Secondary Outcome: Number of Days With Spotting-only in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment.
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 164 | 180
Days | 9.3 (7.5) | 8.6 (5.6)

33. Secondary Outcome: Number of Days With Spotting-only in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 143 | 156
Days | 6.8 (6.2) | 6.4 (4.8)

34. Secondary Outcome: Number of Days With Spotting-only in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 132 | 138
Days | 6.6 (7.1) | 6.3 (4.8)

35. Secondary Outcome: Number of Days With Spotting-only in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 125 | 116
Days | 5.6 (6.1) | 5.6 (3.2)

36. Secondary Outcome: Number of Spotting-only Episodes in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment.
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 164 | 180
Episodes | 1.2 (1.3) | 0.5 (0.8)

37. Secondary Outcome: Number of Spotting-only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 143 | 156
Episodes | 1.0 (1.2) | 0.5 (0.9)

38. Secondary Outcome: Number of Spotting-only Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 132 | 138
Episodes | 0.7 (1.1) | 0.3 (0.6)

39. Secondary Outcome: Number of Spotting-only Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 125 | 116
Episodes | 0.6 (1.1) | 0.2 (0.5)

40. Secondary Outcome: Mean Length of Spotting-only Episodes in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment.
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 97 | 59
Days | 2.64 (1.67) | 2.53 (1.79)

41. Secondary Outcome: Mean Length of Spotting-only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 73 | 48
Days | 2.74 (1.57) | 2.77 (2.24)

42. Secondary Outcome: Mean Length of Spotting-only Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 51 | 26
Days | 2.75 (1.49) | 2.44 (1.54)

43. Secondary Outcome: Mean Length of Spotting-only Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 49 | 21
Days | 2.77 (1.77) | 2.10 (1.27)

44. Secondary Outcome: Maximum Length of Spotting-only Episodes in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment.
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 97 | 59
Days | 3.3 (2.4) | 2.8 (1.9)

45. Secondary Outcome: Maximum Length of Spotting-only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 73 | 48
Days | 3.2 (1.9) | 3.1 (2.4)

46. Secondary Outcome: Maximum Length of Spotting-only Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 51 | 26
Days | 3.5 (2.2) | 2.8 (1.9)

47. Secondary Outcome: Maximum Length of Spotting-only Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 49 | 21
Days | 3.2 (2.3) | 2.2 (1.3)

48. Secondary Outcome: Difference in Duration Between Longest and Shortest Spotting-only Episodes in Reference Period 1
Description: as for outcome 12
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 97 | 59
Days | 1.2 (2.1) | 0.5 (1.1)

49. Secondary Outcome: Difference in Duration Between Longest and Shortest Spotting-only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 73 | 48
Days | 1.0 (1.5) | 0.7 (1.3)

50. Secondary Outcome: Difference in Duration Between Longest and Shortest Spotting-only Episodes in Reference Period 3
Description: Reference Period 3 is defined as Day 181 to Day 270 during study treatment.
Time Frame: From Day 181 to Day 270
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 51 | 26
Days | 1.4 (2.1) | 0.6 (1.6)

51. Secondary Outcome: Difference in Duration Between Longest and Shortest Spotting-only Episodes in Reference Period 4
Description: Reference Period 4 is defined as Day 271 to Day 360 during study treatment.
Time Frame: From Day 271 to Day 360
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 49 | 21
Days | 0.9 (1.9) | 0.2 (0.5)

52. Secondary Outcome: Percentage of Participants With / Without Withdrawal Bleeding at Cycle 1
Description: Withdrawal bleeding is bleeding that occurs when using oral contraceptives (OCs) caused by falling levels and/or taking away external source of estrogen and progestogen toward cycle end.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 180 | 188
Percentage of participants
  without withdrawal bleeding | 25.0 | 12.8
  with withdrawal bleeding | 75.0 | 87.2

53. Secondary Outcome: Percentage of Participants With / Without Withdrawal Bleeding at Cycle 3
Description: as for outcome 52
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 167 | 182
Percentage of participants
  without withdrawal bleeding | 21.0 | 7.7
  with withdrawal bleeding | 79.0 | 92.3

54. Secondary Outcome: Percentage of Participants With / Without Withdrawal Bleeding at Cycle 6
Description: as for outcome 52
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 157
Percentage of participants
  without withdrawal bleeding | 17.7 | 8.3
  with withdrawal bleeding | 82.3 | 91.7

55. Secondary Outcome: Percentage of Participants With / Without Withdrawal Bleeding at Cycle 13
Description: as for outcome 52
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 110 | 110
Percentage of participants
  without withdrawal bleeding | 58.2 | 19.1
  with withdrawal bleeding | 41.8 | 80.9

56. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 1
Description: as for outcome 52
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 135 | 164
Days | 4.2 (2.3) | 6.0 (2.6)

57. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 52
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 132 | 168
Days | 4.3 (2.1) | 5.8 (2.0)

58. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 6
Description: as for outcome 52
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 121 | 144
Days | 4.6 (3.2) | 5.7 (1.9)

59. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 13
Description: as for outcome 52
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 46 | 89
Days | 4.8 (1.8) | 5.5 (1.5)

60. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 1
Description: Intensity was scored as 1=none, 2=spotting, 3=light, 4=normal, or 5=heavy.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 135 | 164
Scores on a scale | 3.2 (0.9) | 4.0 (0.8)

61. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 3
Description: Intensity was scored as 1=none, 2=spotting, 3=light, 4=normal, or 5=heavy.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 132 | 168
Scores on a scale | 3.2 (0.9) | 4.2 (0.7)

62. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 6
Description: Intensity was scored as 1=none, 2=spotting, 3=light, 4=normal, or 5=heavy.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 121 | 144
Scores on a scale | 3.4 (0.8) | 4.0 (0.8)

63. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 13
Description: Intensity was scored as 1=none, 2=spotting, 3=light, 4=normal, or 5=heavy.
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 46 | 89
Scores on a scale | 3.5 (0.7) | 4.1 (0.7)

64. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 1
Description: Onset was defined as the number of days between progestogen withdrawal and the first day of the withdrawal bleeding episode (ie, starting on or after Day 25 for EV/DNG and on or after Day 22 for EE/NGM).
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 135 | 164
Days | 4.7 (7.0) | 4.0 (6.7)

65. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 64
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 132 | 168
Days | 4.3 (7.0) | 3.3 (4.7)

66. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 6
Description: as for outcome 64
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 121 | 144
Days | 5.3 (7.7) | 3.1 (5.1)

67. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 13
Description: as for outcome 64
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 46 | 89
Days | 1.1 (2.2) | 2.1 (1.6)

68. Secondary Outcome: Percentage of Participants With Presence or Absence of Intracyclic Bleeding at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 180 | 188
Percentage of participants
  with absence of intracyclic bleeding | 78.3 | 91.5
  without absence of intracyclic bleeding | 21.7 | 8.5

69. Secondary Outcome: Percentage of Participants With Presence or Absence of Intracyclic Bleeding at Cycle 3
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 167 | 182
Percentage of participants
  with absence of intracyclic bleeding | 79.6 | 85.7
  without absence of intracyclic bleeding | 20.4 | 14.3

70. Secondary Outcome: Percentage of Participants With Presence or Absence of Intracyclic Bleeding at Cycle 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 157
Percentage of participants
  with absence of intracyclic bleeding | 81.6 | 80.3
  without absence of intracyclic bleeding | 18.4 | 19.7

71. Secondary Outcome: Percentage of Participants With Presence or Absence of Intracyclic Bleeding at Cycle 13
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 110 | 110
Percentage of participants
  with absence of intracyclic bleeding | 82.7 | 93.6
  without absence of intracyclic bleeding | 17.3 | 6.4

72. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens. (Episode is a set of days with intracyclic bleeding)
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 180 | 188
Episodes | 0.3 (0.5) | 0.1 (0.3)

73. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 3
Description: as for outcome 72
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 167 | 182
Episodes | 0.2 (0.5) | 0.2 (0.5)

74. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 6
Description: as for outcome 72
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 157
Episodes | 0.2 (0.4) | 0.2 (0.5)

75. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 13
Description: as for outcome 72
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 110 | 110
Episodes | 0.2 (0.4) | 0.1 (0.3)

76. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 39 | 16
Days | 6.7 (8.5) | 6.2 (6.2)

77. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 3
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 34 | 26
Days | 6.6 (6.0) | 4.2 (3.9)

78. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 27 | 31
Days | 5.0 (4.9) | 5.2 (5.0)

79. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 13
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 19 | 7
Days | 3.0 (2.2) | 6.0 (5.9)

80. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 180 | 188
Days | 1.5 (4.8) | 0.5 (2.5)

81. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 3
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 167 | 182
Days | 1.4 (3.8) | 0.7 (2.2)

82. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 157
Days | 0.9 (2.9) | 1.1 (3.1)

83. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 13
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 110 | 110
Days | 0.5 (1.5) | 0.4 (2.1)

84. Secondary Outcome: Percentage of Participants by Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens. Intensity was scored as 1=none, 2=spotting, 3=light, 4=normal, or 5=heavy.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 39 | 16
Percentage of participants
  Spotting | 46.2 | 50.0
  Light | 23.1 | 18.8
  Normal | 15.4 | 18.8
  Heavy | 15.4 | 12.5

85. Secondary Outcome: Percentage of Participants by Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 3
Description: as for outcome 84
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 34 | 26
Percentage of participants
  Spotting | 47.1 | 57.7
  Light | 23.5 | 15.4
  Normal | 20.6 | 23.1
  Heavy | 8.8 | 3.8

86. Secondary Outcome: Percentage of Participants by Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 6
Description: as for outcome 84
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 27 | 31
Percentage of participants
  Spotting | 44.4 | 61.3
  Light | 25.9 | 3.2
  Normal | 18.5 | 19.4
  Heavy | 11.1 | 16.1

87. Secondary Outcome: Percentage of Participants by Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 13
Description: as for outcome 84
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 19 | 7
Percentage of participants
  Spotting | 31.6 | 57.1
  Light | 52.6 | 0.0
  Normal | 10.5 | 28.6
  Heavy | 5.3 | 14.3

88. Secondary Outcome: Percentage of Participants With at Least 1 Intracyclic Bleeding Episode at Cycles 2 to 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: Cycles 2 to 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 184 | 195
Percentage of participants
  Yes | 53.8 | 40.5
  No | 46.2 | 59.5

89. Secondary Outcome: Percentage of Participants With at Least 1 Intracyclic Bleeding Episode at Cycles 2 to 13
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: Cycles 2 to 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 184 | 195
Percentage of participants
  Yes | 62.0 | 49.7
  No | 38.0 | 50.3

90. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI)
Description: Change from Baseline to Cycle 6 in PGWBI Questionnaire's assessment of participant's overall sense of well-being or distress. The PGWBI includes 22 items that, apart from combining into a global overall score, are divided into 6 dimensions: anxiety, depressed mood, positive well-being, self-control, health, and vitality. The response format used a 6-grade Likert scale and the change in the normalized PGWBI global score as well as all the sub-domains score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Scores on a scale
  Global score | 0.41 (6.16) | 1.10 (6.96)
  Anxiety | 0.3 (13.9) | 2.8 (16.8)
  Depressed mood | 0.18 (11.10) | -1.04 (13.73)
  Positive well-being | 49.66 (5.99) | 50.29 (6.60)
  Self-control | 0.69 (9.04) | 0.12 (9.17)
  General health | 81.81 (13.94) | 81.12 (13.38)
  Vitality | -0.17 (8.98) | 0.19 (9.55)

91. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Psychological General Well-Being Index (PGWBI)
Description: Change from Baseline to Cycle 13 in PGWBI Questionnaire's assessment of participant's overall sense of well-being or distress. The PGWBI includes 22 items that, apart from combining into a global overall score, are divided into 6 dimensions: anxiety, depressed mood, positive well-being, self-control, health, and vitality. The response format used a 6-grade Likert scale and the change in the normalized PGWBI global score as well as all the sub-domains score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Scores on a scale
  Global score | -0.14 (7.41) | -0.18 (9.08)
  Anxiety | -1.2 (16.6) | -0.8 (20.4)
  Depressed mood | -0.65 (13.18) | -0.98 (15.96)
  Positive well-being | 0.60 (8.13) | 0.38 (8.43)
  Self-control | -0.49 (9.47) | -0.16 (9.19)
  General health | 0.86 (14.46) | 1.35 (16.15)
  Vitality | 0.28 (10.99) | -0.51 (11.22)

92. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Physical Health
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (physical health - 13 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Scores on a scale | 1.13 (14.09) | 3.44 (14.32)

93. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Physical Health
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (physical health - 13 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Scores on a scale | 1.93 (14.37) | 2.13 (15.21)

94. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Participant Feeling
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (participant feeling - 14 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Scores on a scale | 0.12 (9.76) | 2.19 (10.96)

95. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Participant Feeling
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (participant feeling - 14 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Scores on a scale | -0.44 (12.36) | 0.39 (14.35)

96. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Work
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (work - yes or no; if yes, then 4 choices, and 13 items with a scale of 1-5 [very poor, poor, fair, good, very good]). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 118 | 135
Scores on a scale | 0.54 (9.03) | 0.08 (10.87)

97. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Work
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (work - yes or no; if yes, then 4 choices, and 13 items with a scale of 1-5 [very poor, poor, fair, good, very good]). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 105 | 107
Scores on a scale | -1.38 (12.11) | -1.71 (17.07)

98. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Household Duties
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (household duties - yes or no; if yes, then 4 choices, and 10 items with a scale of 1-5 [very poor, poor, fair, good, very good]). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 140 | 153
Scores on a scale | 1.50 (12.16) | 3.08 (14.83)

99. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Household Duties
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (household duties - yes or no; if yes, then 4 choices, and 10 items with a scale of 1-5 [very poor, poor, fair, good, very good]). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 117 | 125
Scores on a scale | -0.66 (14.31) | 2.83 (18.23)

100. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - School/Course Work
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (school / course work - yes or no; if yes, then 4 choices, and 10 items with a scale of 1-5 (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 28 | 35
Scores on a scale | -0.18 (12.84) | 5.13 (17.43)

101. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - School/Course Work
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (school / course work - yes or no; if yes, then 4 choices, and 10 items with a scale of 1-5 (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 19 | 30
Scores on a scale | -1.97 (18.09) | 4.39 (16.40)

102. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Leisure Time Activities
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (leisure time activities - 6 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Scores on a scale | 1.22 (12.0) | 2.77 (14.36)

103. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Leisure Time Activities
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (leisure time activities - 6 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Scores on a scale | 2.72 (14.45) | 2.37 (15.19)

104. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Social Relationship
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (social relationship - 11 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Scores on a scale | -0.30 (11.15) | 0.41 (13.52)

105. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Social Relationship
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (social relationship - 11 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Scores on a scale | 1.01 (12.58) | 1.75 (13.94)

106. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - General Activities
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (general activities - 16 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Scores on a scale | 0.56 (9.83) | 1.27 (10.55)

107. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - General Activities
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (general activities - 16 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Scores on a scale | 0.73 (10.28) | 1.34 (13.03)

108. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Item Satisfaction
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (item satisfaction). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 110 | 129
Scores on a scale | -0.1 (0.7) | 0.1 (0.9)

109. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Item Satisfaction
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (item satisfaction). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 93 | 107
Scores on a scale | 0.0 (0.6) | 0.1 (0.9)

110. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Overall Life Satisfaction and Contentment
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (overall life satisfaction and contentment). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Scores on a scale | -0.1 (0.7) | 0.0 (0.8)

111. Secondary Outcome: Mean Change From Baseline to Cycle 13 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Overall Life Satisfaction and Contentment
Description: Change from Baseline to Cycle 13 in the overall enjoyment and satisfaction experienced during the past week as scored on the Q-LES-Q (overall life satisfaction and contentment). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Scores on a scale | -0.1 (0.8) | 0.0 (0.8)

112. Secondary Outcome: Percentage of Participants With Improvement in the Investigator's Assessment in Clinical Global Impression (CGI) at Cycle 6
Description: CGI is used to collect information regarding the subject's total clinical experience. The assessment scale ranges from 0 to 7: (0=not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse). The scale of 1, 2, and 3 were categorized as improvement.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Percentage of participants
  Very much improved | 21.1 | 20.0
  Much improved | 41.5 | 25.2
  Minimally improved | 27.2 | 33.5

113. Secondary Outcome: Percentage of Participants With Improvement in the Investigator's Assessment in Clinical Global Impression (CGI) at Cycle 13
Description: as for outcome 112
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Percentage of participants
  Very much improved | 37.9 | 20.3
  Much improved | 32.3 | 26.6
  Minimally improved | 15.3 | 27.3

114. Secondary Outcome: Percentage of Participants With Improvement in the Participant's Assessment in Clinical Global Impression (CGI) at Cycle 6
Description: In 1 section of the CGI the subject rates their total improvement and rate of satisfaction with sexuality during treatment. The assessment scale ranges from 0 to 7: (0=not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse). The scale of 1, 2, and 3 were categorized as improvement.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 147 | 155
Percentage of participants
  Very much improved | 25.2 | 11.6
  Much improved | 32.7 | 30.3
  Minimally improved | 29.3 | 32.2

115. Secondary Outcome: Percentage of Participants With Improvement in the Participant's Assessment in Clinical Global Impression (CGI) at Cycle 13
Description: as for outcome 114
Time Frame: At Cycle 13 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 124 | 128
Percentage of participants
  Very much improved | 33.9 | 17.2
  Much improved | 35.5 | 25.0
  Minimally improved | 16.9 | 28.1

116. Other Pre Specified Outcome: Percentage of Participants With no Increase in Rescue Medication and VAS Decrease During Cycle Days 22 to 28 From Baseline to Cycle 6
Description: Rescue medication was standardized intake of 200 mg Ibuprofen tablets. Baseline: 7 days (Day 22) before first menstrual bleeding to Day 28. Treatment: 7 days (Day 22) before withdrawal bleeding of 6th cycle to Day 28 before the same cycle. The visual analog scale (VAS) is a subject-assessed measure of pelvic pain or headache consisting of a 100 mm long straight line, with verbal anchors at either end, representing a continuum of pain intensity. Accordingly, the scale ranges from 0 mm (absence of pain) to 100 mm (unbearable pain), and the change ranges from -100 mm (best) to 100 mm (worst).
Time Frame: Day 22-28 from Baseline to Day 22-28 from Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 191 | 204
Percentage of participants
  15 mm VAS decrease | 68.1 | 54.4
  30 mm VAS decrease | 58.1 | 42.6
  45 mm VAS decrease | 38.2 | 26.0
  25% VAS decrease | 67.0 | 54.4
  50% VAS decrease | 56.0 | 42.2
  75% VAS decrease | 38.2 | 25.5
  Half-SD decrease | 70.2 | 59.8

117. Other Pre Specified Outcome: The Change of Pelvic Pain or Headache as Determined by the Highest Visual Analog Scale (VAS) Values During Cycle Days 22 to 28 From Baseline to Cycle 6
Description: as for outcome 1
Time Frame: Days 22-28 from Baseline to Days 22-28 from Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Number analyzed (Participants) | 141 | 153
mm | 43.60 (29.16) | 34.55 (30.64)

ADVERSE EVENTS:
Groups:
- Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027): Daily oral administration of one capsule BAY86-5027 [estradiol valerate (EV) / dienogest (DNG)] for 26 days, followed by one capsule placebo for 2 days (28 days total per cycle) for 13 treatment cycles(treatment encapsulated)
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ortho Tri-Cyclen Lo
Serious Adverse Events (participants affected / at risk) | 2/191 | 5/204
Other Adverse Events (participants affected / at risk) | 154/191 | 159/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) (N=191) | Ortho Tri-Cyclen Lo (N=204)
Diabetes insipidus (Endocrine disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 2
Speech disorder (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) (N=191) | Ortho Tri-Cyclen Lo (N=204)
Abdominal distension (Gastrointestinal disorders) | 28 | 35
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 27 | 30
Vomiting (Gastrointestinal disorders) | 19 | 9
Swelling (General disorders) | 3 | 5
Seasonal allergy (Immune system disorders) | 2 | 6
Fungal infection (Infections and infestations) | 6 | 5
Influenza (Infections and infestations) | 8 | 4
Nasopharyngitis (Infections and infestations) | 22 | 20
Sinusitis (Infections and infestations) | 13 | 10
Upper respiratory tract infection (Infections and infestations) | 12 | 11
Urinary tract infection (Infections and infestations) | 23 | 10
Vaginitis bacterial (Infections and infestations) | 7 | 8
Vulvovaginal mycotic infection (Infections and infestations) | 4 | 2
Procedural pain (Injury, poisoning and procedural complications) | 5 | 2
Weight increased (Investigations) | 4 | 4
White blood cells urine positive (Investigations) | 5 | 5
Human papilloma virus test positive (Investigations) | 10 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Dizziness (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 56 | 50
Migraine (Nervous system disorders) | 4 | 3
Sinus headache (Nervous system disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 1 | 5
Mood swings (Psychiatric disorders) | 3 | 7
Amenorrhoea (Reproductive system and breast disorders) | 20 | 1
Breast pain (Reproductive system and breast disorders) | 4 | 3
Breast tenderness (Reproductive system and breast disorders) | 23 | 27
Cervical dysplasia (Reproductive system and breast disorders) | 22 | 20
Dysmenorrhoea (Reproductive system and breast disorders) | 18 | 17
Menorrhagia (Reproductive system and breast disorders) | 4 | 5
Menstruation delayed (Reproductive system and breast disorders) | 5 | 3
Metrorrhagia (Reproductive system and breast disorders) | 31 | 25
Pelvic pain (Reproductive system and breast disorders) | 46 | 47
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Acne (Skin and subcutaneous tissue disorders) | 5 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and/or Principal Investigator shall furnish the Sponsor with a copy of any proposed publication material at least sixty (60) days in advance of the date of submission for publication or presentation so that the proposed publication may be edited appropriately to remove any confidential information before publication or the Sponsor shall have sufficient additional time (not to exceed sixty (60) days) to file a patent application for such Confidential Information.